CLINICAL TRIAL: NCT03117452
Title: Evaluation of a Visual Remediation Intervention for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of California, Riverside (Other); Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Judy L. Thompson, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro20160000350; PC 51-16 (Other Grant/Funding Number: New Jersey Health Foundation)
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; visual processing; cognitive training; visual training
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Half of the participants will be randomized to receive the computerized visual training, which will be delivered in small groups over a period of 12-14 weeks, and the other half will be assigned to the control condition, which consists of standard Partial Hospital care without visual training.
Who Masked: Outcomes Assessor
Masking Description: All participants will be assessed on outcomes of interest by trained clinical interviewers who are blind to the treatment condition in which participants are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual training condition (Experimental): Participants in the visual training condition will participate in the visual training (VT) group, during which they will complete computerized visual training that targets low- and mid-level visual processes. Each group will include a maximum of 3 participants and will meet 3 times a week over a period of 12-14 weeks.
  Interventions: Behavioral: Visual Training
- control condition (No Intervention): Participants assigned to the control condition will receive standard Partial Hospital care without visual training.

INTERVENTIONS:
Behavioral: Visual Training — The computerized visual training (VT) program that is being evaluated was developed by Aaron Seitz, who is a co-investigator on this project; it includes 1) ULTIMEYES, which targets broad-based visual functions, including low-level processes (e.g., visual acuity, contrast sensitivity), and 2) visual perceptual organization exercises, which target mid-level visual processes. Both elements of the program also involve higher-level visual functions, such as visual search and visual attention.
  Arms: visual training condition

SUMMARY:
Schizophrenia is a severe psychiatric condition that is associated with significant distress and disability. In addition to cognitive difficulties in domains such as attention, memory, and problem-solving, individuals with schizophrenia can experience visual-processing abnormalities, including impairments in visual acuity, low-contrast stimulus detection, and perceptual organization (i.e., perceiving visual information in an organized "perceptual whole"). These visual impairments are clinically significant, with research indicating that specific visual-processing alterations are significantly related to poorer performance on higher-level cognitive tasks, impaired facial emotion recognition, impaired reading ability, and worse functional outcomes. Despite such findings, very few studies have evaluated the therapeutic potential of interventions that are specifically designed to improve visual processing ("visual remediation") for individuals with schizophrenia. Thus the aim of this study is to evaluate the efficacy of a computerized visual perceptual training program that targets low- and mid-level visual processes to improve visual, cognitive, and emotion-recognition functions in outpatients with schizophrenia through a small randomized controlled trial. The investigators will recruit up to 40 individuals with schizophrenia or schizoaffective disorder who are receiving treatment in Rutgers University Behavioral Health Care (UBHC) Partial Hospital Program; half will be randomized to receive the computerized visual training, which will be delivered in small groups over a period of 12-14 weeks. The specific aims of this study are to collect preliminary data on: 1) the feasibility of participant recruitment and retention, and tolerability of the treatment components of the study; and 2) the efficacy of computerized visual training (VT) to improve low- and mid-level visual processes, and higher-level cognitive and social-cognitive performance. Based on preliminary data, the investigators hypothesize that the target number of participants will be successfully recruited and engaged in the VT intervention (n=16) and control condition (n=16), and that the participants who receive VT will demonstrate greater improvements on measures of low- and mid-level visual, higher-level cognitive, and social-cognitive functions compared to those who receive standard partial-hospital care without VT. The results of this initial trial will be used to inform the design and application for funding of a larger-scale investigation of visual remediation for individuals with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-60.
* Meets DSM-5 criteria for schizophrenia, schizoaffective disorder, or schizophreniform disorder.
* Currently attends the Rutgers UBHC Partial Hospital Program and plans to continue attending for at least the next 16 weeks.
* If the participant is treated with antipsychotic medication, he/she is on stable treatment with this medication (i.e. no change in medication type, or substantial change in dose, for at least 4 weeks prior to participating in the study and no anticipated change for the next 16 weeks).
* Has capacity to provide informed consent.
* Is fluent in English.
* Has a minimum binocular visual acuity of 20/100, as assessed at baseline using a standard eye chart, with the participant's typical vision correction (e.g., with glasses if the participant typically wears glasses).

Exclusion Criteria:

* Has met DSM-5 criteria for a substance-use disorder within the last 12 months (with the exception of tobacco use disorder, which will be permitted).
* Has a verbal IQ score of < 70 per the Wechsler Test of Adult Reading (WTAR).
* Current or recent history of a medical condition that significantly affects the structure or function of the brain or eye (e.g., ocular or retinal disease, thyroid disease, untreated hypertension, uncontrolled diabetes).
* Current or past neurological or neurodevelopmental disorder such as seizure disorder, cerebral palsy, intellectual disability, or pervasive developmental disorder.
* Has a "lazy eye" or history of severe eye injury.
* Has received electroconvulsive therapy within the last 8 weeks.
* Has a history of head injury with loss of consciousness lasting more than 10 minutes or with neurobehavioral consequences of the injury (e.g., need for follow-up treatment, cognitive or behavioral changes following the injury, etc.).
* Any current use (last month) of non-prescribed amphetamines, opiates, cocaine, sedative-hypnotics, and/or cannabis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
contrast sensitivity | approximately 14 weeks (baseline and post-treatment)
  A measure of low-contrast stimulus detection; contrast sensitivity thresholds at varying spatial frequencies will be examined.
contour integration | approximately 14 weeks (baseline and post-treatment)
  A measure of visual perceptual organization; total number correct, adjusted for guessing, will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Judy L. Thompson, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University Behavioral Health Care (UBHC), Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No